CLINICAL TRIAL: NCT00349804
Title: Intermittent Cold and Dry Air Underneath Football Shoulder Pads as a Method to Assist in Temperature Homeostasis: Evaluation of Efficacy
Brief Title: Intermittent Cold and Dry Air Underneath Football Shoulder Pads
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: NFL Charities (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111-2006
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Body Temperature Regulation
Keywords: temperature; Temperature Homeostasis

ARMS (1):
- Air cooled (COOL) (Other): Subjects will complete the intermitent exercise protocol with cool dry air blown under the shoulder pads during the rest periods and recovery session
  Interventions: Other: cool dry air

INTERVENTIONS:
Other: cool dry air — cool dry air (0.22-0.28 m3/min at 15-18 Degrees C)

SUMMARY:
The purpose of this study is to test if temperature homeostasis in football players can be improved by circulating cool, dry air underneath shoulder pads between periods of intense physical activity.

DETAILED DESCRIPTION:
The purpose of this study is to test if temperature homeostasis in football players can be improved by circulating cool, dry air underneath shoulder pads between periods of intense physical activity. To assess the efficacy of this intervention, several dependent variables will be tested: core body temperature, skin temperature, infrared skin temperature, heart rate, sweating rate, urine color, urine specific gravity, physiological strain index, visual analog thirst, rate of perceived exertion, thermal sensation scale, and fluid intake. The two independent variables (test variables) are treatment which has two levels (Control - no air blown under the shoulder pads, COOL - cool, dry air blown under the shoulder pads) and time (pre-exercise and post-exercise cycles, rest break and recovery).

Specific Aim 1: To assess differences in physiological parameters when cooled dry air is blown under football shoulder pads as a means of cooling football players between periods of exercise and after exercise. Limited research is available to demonstrate the efficacy of cooling methods alternated with vigorous exercise. Football players are at particular risk for heat-related illness because they frequently practice and compete in hot, humid conditions in uniforms that limit the body's natural thermoregulation. To study this specific aim, three hypotheses will be addressed during the data collection process of this investigation: (1) a significantly lower increase in core body temperature, heart rate, skin temperature, and infrared skin temperature will be noted during the COOL testing sessions as compared to the Control sessions; (2) significantly lower measurements of urine color, urine specific gravity, and sweat rate will be noted in the COOL testing sessions as compared to the Control sessions; and (3) significant associations will be noted between core body temperature and infrared temperature during both testing sessions.

Specific Aim 2: To assess differences in subjective ratings of exertion and heat stress during and after exercise sessions when cooled dry air is blown under football shoulder pads as compared to no air during rest breaks between the exercise bouts. The rationale behind Specific Aim 2 is that the cooling method (COOL) will aid in improving the body's blunted cooling mechanisms. The sensation of the cool, dry air will be more prominent than the sensation of warmth (during the COOL trials), the decrease in physiological strain, and the decrease in core body temperature will cause the subject to experience lower perceived exertion; thus, subjects' subjective response to exertion in subsequent exercise cycles will be decreased. One hypothesis will be addressed related to this specific aim: cool, dry air blown under football shoulder pads (COOL) as a cooling method between exercise bouts will significantly lower physiological strain index score, visual analog thirst score, rate of perceived exertion, and thermal sensation score as compared to no cool, dry air being blown under the shoulder pads (Control).

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* ages 18-30 years

Exclusion Criteria:

* a health questionnaire to identify any contraindications will be given during screening

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Heart rate | (baseline, min 25, min 50 and post (min 75))
Physiological strain index (PSI) | (baseline, min 25, min 50 and post (min 75))
Visual analog thirst scale (VATS) | (baseline, min 25, min 50 and post (min 75))
Rate of perceived exertion (RPE) | (baseline, min 25, min 50 and post (min 75))
Thermal sensation scale (TSS) | (baseline, min 25, min 50 and post (min 75))

SECONDARY OUTCOMES:
Fluid intake during trials | Post measurement (total consumed)
Urine color | (pre and post)
Specific gravity | (pre and post)

CONTACTS AND LOCATIONS:
Overall Officials: MaryBeth Horodyski, EdD, ATC, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States